CLINICAL TRIAL: NCT01072864
Title: Effects of California Walnuts on Vascular Function in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Robert M. Hackman, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200917508-1
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Cardiovascular Diseases
Keywords: Postmenopausal
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 g of walnuts (Experimental)
  Interventions: Other: Walnuts
- 20 g of walnuts (Experimental)
  Interventions: Other: Walnuts
- 30 g of walnuts (Experimental)
  Interventions: Other: Walnuts
- 40 g of walnuts (Experimental)
  Interventions: Other: Walnuts

INTERVENTIONS:
Other: Walnuts — Consumption of 5 g of walnuts.
  Arms: 5 g of walnuts
Other: Walnuts — Consumption of 20 g of walnuts.
  Arms: 20 g of walnuts
Other: Walnuts — Consumption of 30 g of walnuts.
  Arms: 30 g of walnuts
Other: Walnuts — Consumption of 40 g of walnuts.
  Arms: 40 g of walnuts

SUMMARY:
To determine the potential acute cardiovascular benefits of California Walnuts in postmenopausal women of ages 55-70.

Primary outcome measures:

* Vascular function
* Platelet reactivity

We hypothesize that the consumption of California walnuts will improve vascular function and platelet reactivity.

DETAILED DESCRIPTION:
Epidemiological studies have shown that consumption of high amounts of plant foods, such as nuts, fruits and vegetables, appears to be protective against chronic diseases including heart disease, stroke, diabetes mellitus and metabolic syndrome. In recent years, numerous studies indicate that consumption of walnuts mainly containing α-linolenic acid (ALA), L-arginine and polyphenols beneficially alters vascular function and reduces inflammatory biomarkers. Recent studies have reported that consumption of walnuts is associated with beneficial effects in prevention of chronic diseases by favorably altering human serum profiles (i.e. decrease in LDL cholesterol and triglycerides and increase in HDL cholesterol and apolipoprotein A1) which are closely involved in the development of cardiovascular disease (CVD). In addition, recent reports by Dr. Ros and his colleagues indicate that addition of walnuts to a high-fat meal can improve endothelial function. This favorable influence on vasoactivity has been attributed to the antioxidant and anti-inflammatory properties of components of walnuts.

Due to their age and menopausal status, postmenopausal women in particular, are at a greater risk population for developing CVD. Males tend to show greater rates of CVD than pre-menopausal women, while women following menopause show an increase in the rates of CVD. This increase is associated with endothelial dysfunction and decreased vasodilation which are apparently expressed after menopause and become worse with age. In this study, we will define the effects of consuming California walnuts on vascular health.

We hypothesize that consumption of California walnuts, which are particularly rich in ALA, L-arginine and polyphenols, will improve endothelial function and platelet reactivity in an at-risk population of postmenopausal women 50-70 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years of age
* Lack of menses in the last year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing to consume up to 40 g of California walnuts.
* BMI 18.5-34.9 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Weight <110 pounds
* Diabetes
* Taking anticoagulation medication including NSAIDs
* Blood pressure ≥ 160/90 mm Hg
* PFA-100 readings 10 % outside of normal reference range (normal reference range for ADP-Collagen: 71-118 sec; Epinephrine-Collagen: 94-193 sec).
* Renal or liver disease
* Heart disease, which includes cardiovascular events and Stroke
* Cushing's syndrome
* Chronic/routine high intensity exercise
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or CMP (laboratory values outside the reference range) if determined to be clinically significant.
* History of cancer
* History of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year.
* Use of MAOI inhibitor within the last 1 year (e.g. phenelzine (Nardil), tranylcypromine (Parnate), etc)
* Malabsorption
* Anxiety medications
* Routine use of prescription drugs or over-the counter medications, which may potentially modulate the outcome of this study; including antibiotics, aspirin and aspirin-containing formulations, COX-2 inhibitors, antihistamines, corticosteroids, ACE-inhibitors, and beta-blockers.
* Asthma (can be worsened by mild to moderate food allergies).
* Indications of substance or alcohol abuse within the last 3 years
* Use of multivitamin/mineral supplements
* Use of herbal or plant-based supplements; omega-3 fatty acids, and fish oils in the past 3-6 months.
* Nut allergies
* Soy-derived supplements
* Soy/soy products consumption > 2 servings/week
* Hormone replacement therapy
* Alcohol consumption > 1 drink/day (i.e. 1 bottle of beer, ½ glass of wine, and 1 shot of hard liquor)
* Fruit consumption ≥ 3 cups (6 servings)/day
* Vegetable consumption ≥ 4 cups (8 servings)/day
* Grain consumption ≥ 8 oz/day
* Meat and Beans ≥ 7 oz/day
* Fatty Fish ≥ 3 times/week
* Milk ≥ 5 cups/day
* Oil ≥ 8 tsp/day
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry (PAT) | 2 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Hackman, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States